CLINICAL TRIAL: NCT03365817
Title: Cognitive Function and Addiction in Patients With Chronic Pain Under Opioid Tapering in a Multidisciplinary Pain Treatment
Brief Title: Cognitive Function and Addiction Under Opioid Tapering
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Hørslev-Fonden (Unknown)
Responsible Party: Principal Investigator, Per Sjogren, Professor in palliative Medicine, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-B-2008-061
Record Dates: First submitted 2017-11-22; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pain; Opioid Use
Keywords: cognitive function; opioid dependence; opioid withdrawal; quality of life; side effect
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders | interventions — Morphine; Oxycodone; Fentanyl; Tramadol

STUDY DESIGN:
Intervention Model Description: Random assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taper off (Experimental): Decrease of opioid daily dose until discontinuation for up to six months.
  Interventions: Drug: Opioids taper off
- Control Group (Active Comparator): No changes on opioids and adjuvant medication for up to six months.
  Interventions: Drug: Opioid stable treatment

INTERVENTIONS:
Drug: Opioids taper off — Decrease of 10% of opioid daily dose every one to two weeks until discontinuation for up to six months.
  Other Names: Morphine, oxycodone, metadone, fentanyl, tramadol
  Arms: Taper off
Drug: Opioid stable treatment — No changes on prescribed opioids and adjuvant medication for the next six months
  Arms: Control Group

SUMMARY:
This study evaluates the effects of opioid dose reduction in the treatment of chronic pain in adults. Participants were divided in two groups: 1) patients that reduced opioid dose and 2) patients that kept the same opioid dose for six months.

DETAILED DESCRIPTION:
BACKGROUND The indications for initiating long-term opioid treatment for chronic non-cancer pain are often unclear and may be associated with poor outcomes and problematic use. Few available studies demonstrated that opioids do not provide advantages regarding pain control, quality of life and functional capacity in this population and may have numerous serious adverse effects and consequences.

AIMS

This study aimed at:

1. evaluating the feasibility of a opioid tapering off program to patients with chronic pain,
2. investigating the influence of opioid tapering off on cognitive function, pain, symptoms of opioid withdrawal, anxiety , depression, and health related quality of life,
3. investigating the prevalence of addiction in chronic pain patients in a long-term treatment,
4. determining the predictive value of the Pain Medication Questionnaire (PMQ) in patients with chronic pain,
5. investigating how opioid tapering off influences PMQ.

METHODS

Study design

This is a prospective, single centre, open-label, parallel-group randomized controlled trial (1:1) conducted at the Multidisciplinary Pain Centre of Rigshospitalet, Copenhagen University Hospital, Denmark.

Two phases with nine assessments were planned. The Phase 1 was the stabilization phase and consisted of two assessments: the first assessment (baseline) was done when patients were admitted to the pain centre and the second assessment was done when medical treatment was considered stable for at least three weeks (stable dose levels and regular intervals). In the following patients went through Phase 2 and were randomized to receive the intervention (Taper off Group) or continue the same stable treatment (Control Group). Seven assessments were planned to this phase: third and fourth assessments were done in intervals of two to three weeks and the following assessments (fifth to ninth) with intervals of one month in between.

Intervention

The taper-off intervention consisted of a reduction of 10% of the daily opioid dose every 1-2 weeks until discontinuation of opioid treatment for up to six months. Clonidine use (25mg - 150mg/day) was allowed in cases of opioid withdrawal symptoms, according to medical prescription.

Analysis

Statistical analysis will be performed to compare baseline characteristics between groups (patients that complete the study vs. patients that dropped out and intervention vs. control group). Comparative analysis of primary and secondary outcomes between groups will also be performed to identify significant differences associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old or more
* at least seven years of schooling
* pain duration of at least six months,
* treatment with oral opioids for more than three months
* daily opioid dose ≥ 60 mg of oral morphine equivalent

Exclusion Criteria:

* not fluent in Danish language
* cancer disease
* poor general health condition
* pregnancy, dementia
* encephalopathy
* brain damage
* cranial base trauma
* enrolled in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Cognitive function - sustained attention | Through study completion up to 4 years.
  EKHO, computer program that registers the continuous reaction time to respond to the emission of a sound signal. Scores were summarized in milliseconds using 10th (fastest values), 50th and 90th (slowest values) percentiles. More prolonged times mean worse performance.
Cognitive function - psychomotor speed | Through study completion up to 4 years.
  Finger Tapping Test, a mechanical device with a key attached was used to record the number of taps. Score was calculated by the numbers of taps, considering the average of each hand and the differences between hands. Higher scores mean better performance.
Cognitive function - working memory | Through study completion up to 4 years.
  Digit Span Test, subjects should repeat orally series of numbers of increasing lengths, in forward and backward orders. Scores were calculated separately for forward and backward exercises, considering the number of correct repetitions. Scores range from 0 to 14. Higher scores mean better performance.
Cognitive function - mental flexibility | Through study completion up to 4 years
  Trail Making Test B, numbers and letters written on a paper should be connected in alternated sequence and increasing order. Score was calculated by the total time spent to correctly conclude the test (seconds). Shorter time mean better performance.
Cognitive function - mental state | Through study completion up to 4 years.
  Mini Mental State Examination, measures orientation to time and place, registration of words, attention, calculation, and word recall, as well as language and visual construction. Total scores range from 0 to 30; scores below 27 were considered indicative of cognitive dysfunction.
Risk of opioid misuse | Through study completion up to 4 years.
  Pain Medication Questionnaire, 26 items responded on a 5-point Likert format scale. Scores range from 0 to 104, higher score means higher risk of opioid misuse. Scores equal or above 22 were considered indicative of risk for opioid addiction.

SECONDARY OUTCOMES:
Pain intensity | Through study completion up to 4 years.
  Verbal numerical scale from 0=no pain to 10= worst pain, to assess pain right now and average pain.
Sleep | Through study completion up to 4 years.
  Number of total hours of sleep in the previous night before assessment
Rest | Through study completion up to 4 years.
  Rest sensation assessed by the question "do you feel rested?". Answers were categorized as yes or no.
Quality of life | Through study completion up to 4 years.
  RAND 36-Item Short Form Health Survey version 1.0., 36 items distributed in 8 scales: physical functioning, bodily pain, role limitations due to physical health, role limitations due to emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item was scored on a 0 to 100 range. Items in the same scale were averaged together to create the 8 scale scores. A high score defines a more favorable health state.
Depression and anxiety | Through study completion up to 4 years.
  Hospital Anxiety and Depression Scale, self-assessment about the last week. It has 14 items divided in anxiety subscale and depression subscale with seven items each one.The maximum score for each scale is 21; cut-off scores for each scale were 8 to 10 for possible and 11 or higher for probable presence of mood disorder.
  A clinical judgment was also done by the pain specialist physician (possible answers were yes or no)
Objective symptoms of opioid withdrawal | Through study completion up to 4 years.
  Objective Opiate Withdrawal Scale, 13 physically observable signs, rated present or absent that reflected common motoric and autonomic manifestations of opiate withdrawal: yawning, rhinorrhea, piloerection, perspiration, lacrimation, mydriasis, hands tremors, hot and cold flashes (shivering), restlessness (frequent shifts of position), vomiting. muscle twitches, abdominal cramps, and anxiety. Scores range from 0 to 13, higher scores mean more opioid withdrawal symptoms.
Subjective symptoms of opioid withdrawal | Through study completion up to 4 years.
  Subjective Opiate Withdrawal Scale, self-assessment, 16 items: motoric, autonomic, gastrointestinal, and musculoskeletal opiate withdrawal symptoms and indirectly related psychological symptoms, like anxiety and craving. Answers are scored from 0 to 4 based on how patient is feeling at the time of assessment. Scores range is 0-64, higher scores mean more opioid withdrawal symptoms.
Addiction - Portnoy's Criteria | Through study completion up to 4 years.
  Classification according to Portnoy's Criteria (psychological dependence, evidence of compulsive drug use, and evidence of a group of associated behaviors). Subjects were classified in addict and non-addict.
Addiction - International Classification of Diseases -10. | Through study completion up to 4 years.
  Diagnostic criteria according to the International Classification of Diseases -10. Subjects should present at least three symptoms associated with addiction in the least month or several times within a year to be considered addict.

CONTACTS AND LOCATIONS:
Overall Officials: Per Sjøgren, DMSc, Principal Investigator — Rigshospitalet, Denmark; Jette Højsted, MD, Principal Investigator — Rigshospitalet, Denmark